CLINICAL TRIAL: NCT06696664
Title: Exploring the Genome-wide Association Study of the Advantageous Population for Clinical Cure of Chronic Hepatitis B With Long-acting Interferon Therapy
Brief Title: Exploring the Genome-wide Association Study of the Population With Clinical Cure Advantage in the Treatment of Chronic Hepatitis B With Long-acting Interferon
Status: Recruiting | Type: Observational
Sponsor: Minghui Li (Other Government)
Responsible Party: Sponsor-Investigator, Minghui Li, Director and Professor, Beijing Municipal Administration of Hospitals
Organization: Beijing Municipal Administration of Hospitals (Other Government)
Other Study IDs: BTP-CHB04
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; pegylated interferon-α; clinical cure; gene sequencing; genetic polymorphism
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 96 Weeks
Biospecimen Retention: Samples With DNA — Collect blood samples as candidate gene sequencing samples, use high-throughput sequencing technology to detect the whole genome of the subjects, identify relevant gene loci that have predictive value for clinical cure of chronic hepatitis B treated with PEG-IFN - α, and establish a predictive model and calculation formula between gene polymorphism and the efficacy of PEG-IFN - α antiviral therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Case group (HBsAg negative conversion group): 120 CHB patients who achieved clinical cure after continuous treatment with PEG-IFN-α for more than 24 weeks.
  Interventions: Drug: PEG-IFN-α
- Control group: Control group: 300 CHB patients who were continuously treated with PEG-IFN - α for more than 24 weeks without clinical cure.
  Interventions: Drug: PEG-IFN-α

INTERVENTIONS:
Drug: PEG-IFN-α — chronic hepatitis B (CHB) who were continuously treated with pegylated interferon (PEG-IFN - α) for more than 24 weeks

SUMMARY:
This study is a real-world case-control study conducted, with 120 CHB patients who received continuous treatment with PEG-IFN-α for more than 24 weeks as study subjects. Among them, the clinical cure group obtained through PEG-IFN-α treatment is the case group; The group that did not achieve clinical cure after PEG-IFN-α treatment was used as the control group, and the case group and control group were allocated cases in a 2:1 ratio. Collect blood samples from subjects as sequencing samples for candidate genes, use high-throughput sequencing technology to detect the whole genome of subjects, identify relevant genetic polymorphism that have predictive value for clinical cure of chronic hepatitis B treated with PEG-IFN-α, and establish a predictive model and calculation formula between gene polymorphism and the efficacy of PEG-IFN-α antiviral therapy.

DETAILED DESCRIPTION:
This study is a real-world case-control study conducted on 120 patients with chronic hepatitis B (CHB) who were continuously treated with pegylated interferon-α (PEG-IFN-α) for more than 24 weeks. Among them, the clinical cure group obtained through PEG-IFN-α treatment is the case group; The group that did not achieve clinical cure after PEG-IFN-α treatment was used as the control group, and the case group and control group were allocated cases in a 2:1 ratio. Collect blood samples as candidate gene sequencing samples, use high-throughput sequencing technology to detect the whole genome of the subjects, identify relevant genetic polymorphism that have predictive value for clinical cure of chronic hepatitis B with PEG-IFN-α therapy, and establish a predictive model and calculation formula between gene polymorphism and the efficacy of PEG-IFN-α antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤ 70 years old, Han ethnicity, gender not limited;
* According to the "Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2022)", patients with HBsAg and/or HBV DNA positivity for more than 6 months and chronic inflammatory liver disease caused by persistent HBV infection are diagnosed with chronic hepatitis B (CHB);
* The patient receives subcutaneous injections of PEG-IFN-α for at least 24 consecutive weeks;
* Patients voluntarily sign an informed consent form before the start of the study.

Exclusion Criteria:

* Patients with co infection of HCV, HDV, HIV, and Treponema pallidum;
* Patients with evidence of alcohol abuse, decompensated cirrhosis, liver tumors (liver cancer or AFP>100 ng/ml), or autoimmune diseases.
* Patients who become pregnant during PEG-IFN - α treatment;
* Other situations that the patient deems unsuitable for inclusion in this trial.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Collect blood samples from CHB patients who have completed PEG-IFN - α continuous treatment for more than 24 weeks (two groups of CHB patients who have obtained and have not obtained clinical cure after PEG-IFN - α treatment), to provide samples for sequencing candidate genes.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical cure | 96 weeks
  HBsAg negative, with or without the presence of anti HBs, HBV DNA below the lower limit of detection, ALT<lower limit of normal value
Non clinical cure | 96 weeks
  Non clinical cure (partially effective and ineffective): HBsAg has not turned negative Partially effective: HBV DNA is below the lower limit of detection, ALT is below the lower limit of normal. Invalid: Not partially valid.

SECONDARY OUTCOMES:
HBV DNA turns negative | 96 weeks
  HBV DNA suppression (HBV DNA below the detection limit or not detected);
HBeAg conversion to negative | 96 weeks
  HBeAg conversion to negative (disappearance of HBeAg in patients with previous HBeAg positivity).
HBsAg re positivity rate | 96 weeks
  Hepatitis B surface antigen re positive rate after PEG-IFN-α withdrawal
Improvement in liver function | 96 weeks
  Liver function status after PEG-IFN-α treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No